CLINICAL TRIAL: NCT04292249
Title: Predictive Value of suPAR and hsCRP on Postoperative Mortality in 951 Patients Undergoing Elective On-pump Cardiac Surgery
Brief Title: Predictive Value of suPAR and hsCRP on Postoperative Mortality in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Persimune (Unknown); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Sebastian Roed Rasmussen, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: H-18002379
Record Dates: First submitted 2020-02-24; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Thoracic Surgery; Cardiac Surgical Procedures; Biomarkers
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples:
  The blood samples for the study were drawn preoperatively or within 24 hours of surgery and stored in the Persimune Biobank or two other biobanks at Dept. Cardiothoracic Anaesthesiology and Dept. Cardiothoracic Surgery, Rigshospitalet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elective on-pump cardiac surgery patients: Adult patients (≥18 years) undergoing elective on-pump cardiac surgery (isolated coronary artery bypass graft (CABG), single and multiple valvular procedures, combined CABG and valvular surgery, and others).
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Analysis will be performed using commercially available analyses (suPARnostic® kit (validated to measure suPAR concentrations between 0.6 and 22 ng/mL) (ViroGates)). HsCRP will be measured by high sensitivity CRP assays (Tina-quant hs-CRP latex assay (validated to measure CRP concentrations between 0.3 - 20 mg/L) (Roche/Hitachi)). In patients with CRP>20 mg/L a regular CRP-measurement will be performed.

SUMMARY:
This study aims to investigate whether preoperative soluble urokinase plasminogen activating receptor (suPAR) and High-sensitivity C-Reactive Protein (hsCRP) are independent markers of death after cardiac surgery. Further, to assess whether suPAR and hsCRP provides increased predictive accuracy of the clinical risk model EuroSCORE II. The purpose of the study is to gain knowledge on whether these inflammatory biomarkers might be able to reveal a pro-inflammatory disease state that represents a significant risk in patients undergoing cardiovascular surgery. Hence, these biomarkers may assist clinicians in selecting compassionate treatment for high risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Planned elective on-pump cardiac surgery (isolated coronary artery bypass graft (CABG), single and multiple valvular procedures, combined CABG and valvular surgery, and others)
* Given informed consent on delivering a blood sample for the biobank.

Exclusion Criteria:

* Peroperatively cancelling the surgery
* Sudden change to off-pump coronary artery bypass (OPCAB) surgery
* Death prior to surgery
* Project blood samples not available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) undergoing cardiac surgery at department of Cardiothoracic Surgery at Rigshospitalet, Copenhagen University Hospital, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 951 (Actual)
Dates: Start 2012-08-06 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Association of preoperative suPAR values in relation to the censored time-to-event outcome "death from any cause" | from index surgery to censoring date 12.31.2018

SECONDARY OUTCOMES:
Association of preoperative hsCRP values in relation to the censored time-to-event outcome "death from any cause" | from index surgery to censoring date 12.31.2018
Assess whether adding suPAR, hsCRP or combined suPAR+hsCRP measurements improves predictive accuracy of EuroSCORE II | from index surgery to 30 days postoperative
Sensitivity of the models; EuroSCORE II, suPAR, hsCRP, suPAR+hsCRP, EuroSCOREII+suPAR, EuroSCOREII+hsCRP and EuroSCOREII+suPAR+hsCRP in relation to the time-to-event outcome "death from any cause" | from index surgery to 30 days postoperative
Specificity of the models; EuroSCORE II, suPAR, hsCRP, suPAR+hsCRP, EuroSCOREII+suPAR, EuroSCOREII+hsCRP and EuroSCOREII+suPAR+hsCRP in relation to the time-to-event outcome "death from any cause" | from index surgery to 30 days postoperative

OTHER OUTCOMES:
30 days mortality measured by a yes/no question of "all-cause mortality" | from index surgery to 30 days
1-year mortality measured by a yes/no question of "all-cause mortality" | from index surgery to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian R Rasmussen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Cardiothoracic Anaesthesiology, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT04292249/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT04292249/SAP_001.pdf